CLINICAL TRIAL: NCT03591640
Title: The Validity of Kleinhauer Betke in Women With Known Hemoglobinopathy for Fetal-maternal Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HYMC-0057-18
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Fetal-Maternal Hemorrhage
MeSH Terms: conditions — Fetomaternal Transfusion | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant with hemoglobinopathy (Active Comparator): Standard of care with blood test before active labor
  Interventions: Diagnostic Test: Blood test
- Pregnant without known hemoglobinopathy (Active Comparator): Standard of care with blood test before active labor
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — Standard blood test

SUMMARY:
The aim of this study is to determine the validity of Kleinhauer Betke in women with known hemoglobinopathy for fetal-maternal hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant with singleton fetus
* Gestational age 34-42
* With or without known hemoglobinopathy

Exclusion Criteria:

* Known risk factor for fetal maternal hemorrhage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 27 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Validity of Kleinhauer Betke test in Pregnant Women | 24 hours
  Comparison of Kleinhauer Betke results with electrophoresis results to determine presence of F-hemoglobin. This would indicate the validity of the Kleinhauer Betke test in women with hemoglobinopathy

CONTACTS AND LOCATIONS:
Overall Officials: Rinat Gabbay-Benziv, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No